CLINICAL TRIAL: NCT03295812
Title: Stratification of Chronic Alcoholic Liver Diseases (SCALE Study) Based on Organs Injury: a Multi-center Prospective Observational Study
Brief Title: Stratification of Chronic Alcoholic Liver Diseases (SCALE Study)
Acronym: SCALE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: 004
Record Dates: First submitted 2017-09-25; First posted 2017-09-28 (Actual); Last update posted 2018-01-23 (Actual); Status verified 2017-09

CONDITIONS: Alcoholic Liver Disease
MeSH Terms: conditions — Liver Diseases, Alcoholic | interventions — Standard of Care

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma, serum, urine and DNA samples will be reserved
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: standard therapy — standard therapy,non-interventional study

SUMMARY:
Recent years, the European Association for the Study of the Liver-chronic liver failure (EASL-CLIF) has defined and graded acute-on-chronic liver failure (ACLF) based on CANONIC study which enrolled cirrhotic patients with acute decompensation. However, the characteristics and definitions of ACLF in non-cirrhotic patients with acute deterioration of liver function and organs injury or failure remain to be clear. As for patients who don't fulfil ACLF criteria, there might be a subgroup with high risk of progression (>25%) and a moderate 4-week mortality rate (>7%), which can be defined as "pre-ACLF", while the others are just chronic liver disease with "mere" liver injury or decompensation. This stratification system was primarily verified in a previous retrospective cohort which enrolled Hepatitis B patients only. The stratification criteria for chronic alcoholic liver disease needs to be further defined in detail. Therefore, investigators plan to prospectively recruit 3000 chronic alcoholic hospitalized patients with liver dysfunction from 24 hepatology departments in China, aiming to propose a stratified diagnostic system for chronic alcoholic patients based on organs injury. Meanwhile, risk factors of disease progression and short-term mortality will be analyzed, while characteristics and prognosis will be compared between patients with and without cirrhosis.

ELIGIBILITY:
Inclusion Criteria:

1. Long-term alcohol consumption (at least one of the followings):

   1. >40g/d for male and >20g/d for female, at least for 5 years;
   2. >50g/d for at least 6 months;
2. Liver injury (at least one of the followings):

   1. AST>1.0 ULN and AST>ALT;
   2. TBIL>2.0mg/dl;
   3. Ascites;
   4. Hepatic encephalopathy;
   5. Esophageal variceal bleeding;
   6. Hypersplenism

Exclusion Criteria:

1. Younger than 18 or older than 80;
2. Other etiologies rather than alcoholic liver disease, including but not limited to the followings:

   1. Acute or chronic virologic hepatitis: Hepatitis A-E, Hepatitis caused by CMV,EBV, etc.
   2. Autoimmune hepatitis, including PSC, PBC, AIH, IgG4 related liver disease
   3. Inherited metabolic liver diseases: Wilson disease;
   4. Others: Schistosomiasis
3. HIV antibody positive;
4. Malignancies including but not limited to HCC;
5. Pregnancy;
6. Hospital stay less than 24h;
7. Refuse to sigh the informed consent;
8. Combined with other improper situations determined by investigators.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be selected from all in-patients in 24 hepatology departments
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2017-11-16 (Actual); Primary Completion 2019-12-30 (Estimated); Study Completion 2020-12-30 (Estimated)

PRIMARY OUTCOMES:
4-week mortality | 4 weeks
  mortality rate
12-week mortality | 12 weeks
  mortality rate

SECONDARY OUTCOMES:
4-week progression rate | 4 weeks
  The proportion of subjects progressed to acute-on-chronic liver failure within 4 weeks
24-week mortality | 24 weeks
  mortality rate
48-week mortality | 48 weeks
  mortality rate

OTHER OUTCOMES:
Risk factors for disease progression within 4 weeks | 4 weeks
  analysis of risk factors for disease progression

CONTACTS AND LOCATIONS:
Overall Officials: Jinjun Chen, Principal Investigator — Hepatology Unit, Department of Infectious Diseases, Nanfang Hospital, Southern Medical University
Locations (26):
- China (26):
  - Nanfang Hospital, Guangzhou, Guangdong
  - People's hospital of Yangshan, Qingyuan, Guangdong
  - Dongguan dalang hospital, Dongguan
  - People's hospital of Foshan Nanhai District, Foshan
  - The First People's Hospital of Foshan, Foshan
  - Guangdong General Hospital, Guangzhou
  - Guangzhou Eighth People's Hospital, Guangzhou
  - The First Affiliated Hospital,Guangzhou University of Chinese Medicine, Guangzhou
  - The First Affiliated Hospital,Jinan University, Guangzhou
  - Huizhou Central Hospital, Huizhou
  - Huizhou Hospital of Traditional Chinese Medicine, Huizhou
  - The First People's Hospital of Huizhou, Huizhou
  - The Sixth People's Hospital of Huizhou, Huizhou
  - The Third People's hospital of Huizhou, Huizhou
  - People's Hospital of Enping, Jiangmen
  - Kaiping Central Hospital, Kaiping
  - The Second People's Hospital of Yuebei, Shaoguan
  - Peking University Shenzhen Hospital, Shenzhen
  - Shenzhen Third People's Hospital, Shenzhen
  - Shunde Hospital of Southern Medical University, Shunde
  - Yangjiang Public Health Hospital, Yangjiang
  - People's Hospital of Yingde City, Yingde
  - Nongken Central Hospital, Zhanjiang
  - The First People's Hospital of Zhaoqing, Zhaoqing
  - Zhaoqing No.2 People's Hospital, Zhaoqing
  - Zhongshan Second People's Hospital, Zhongshan